CLINICAL TRIAL: NCT00903994
Title: An Open-Label, Phase II, Pilot Study on the Onset of Action of KTP, 20% in the Treatment of Acute Pain Associated With Tendonitis or Bursitis of the Shoulder, Elbow or Knee
Brief Title: A Pilot Study on the Onset of Action of KTP, 20% in the Treatment of Acute Pain Associated With Tendonitis or Bursitis of the Shoulder, Elbow or Knee
Acronym: KTP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Sr. Director Clinical R&D, Endo Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: EN3269-201; Ketoprofen Topical Patch, 20%
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Tendonitis of the Shoulder, Elbow, or Knee
Keywords: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): Single Arm
  Interventions: Drug: Ketoprofen Topical Patch 20%

INTERVENTIONS:
Drug: Ketoprofen Topical Patch 20% — Ketoprofen is a pressure-sensitive adhesive material containing 20% Ketoprofen which is applied to a polyester textile and covered with a foil release liner.for the treatment of mild to moderate acute pain associated with Tendonitis or Bursitis of the shoulder, elbow or knee

SUMMARY:
Open-label study to be conducted at 2 US investigational sites in subjects who have acute tendonitis or bursitis of the shoulder, elbow, or knee. Eligible subjects receive treatment with the KTP, applied once daily at the same application site for 3 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Are males or females 18 years of age or older (If female, must be practicing abstinence or using a medically acceptable form of contraception (e.g., intrauterine device, hormonal birth control, or double barrier method). For the purpose of this study, all females are considered to be of childbearing potential unless they are post-menopausal, biologically sterile, or surgically sterile (i.e., hysterectomy, bilateral oophorectomy), or have undergone tubal ligation for greater than or equal to one year.)
* Have a diagnosis of acute tendonitis or bursitis of the shoulder, elbow or knee with acute onset of the current episode in the 15 days preceding the screening visit
* Have average pain intensity during daily activities over the past 24 hours rated 5 or greater on an 11-point scale (range 0 to 10). (If the onset of acute tendonitis or bursitis is less than 24 hours before the screening visit, the patient will rate the average pain intensity during daily activity since the time of onset.) Site personnel must not reveal this eligibility criterion to prospective patients.
* Are willing to discontinue use of all analgesic medications (including over-the-counter [OTC] analgesics) except the study patch. Note: Aspirin at a daily dose of 81 mg per day for cardiovascular prophylaxis will be allowed.
* Have been informed of the nature of the study and have provided written informed consent

Exclusion Criteria:

* Have a positive urine pregnancy test (females of childbearing potential only) or are pregnant or lactating
* Have tendonitis or bursitis secondary to a systemic inflammatory disease (e.g., rheumatoid arthritis, spondyloarthropathies), or resulting from calcification or requiring surgery
* Have had pharmacologic treatment (e.g., analgesic medications except 81mg prophylactic aspirin) less than 12 hours before the baseline assessments
* Have received systemic corticosteroids in the 30 days preceding the screening visit (e.g., intra-articular, peritendinous, oral, or parenteral administration). Nasal inhalation steroids are permitted.
* Have received any pharmacologic treatment or physical therapy in the past 6 months for the joint targeted for this study. Pharmacologic treatment or physical therapy for current tendonitis or bursitis is allowed unless the medication or therapy is prohibited by the protocol.
* Require continued use of an immobilization device for treatment of the current episode of tendonitis or bursitis
* Have a history or physical examination finding that is incompatible with safe participation in the study, including GI ulcer or bleeding, anemia or prolonged bleeding time
* Have a history, or physical examination finding, that is incompatible with study product use or with obtaining robustly interpretable data, chronic skin conditions such as psoriasis, clinically significant osteoarthritis, or skin lesions or wounds at the affected site
* Have a history of drug or alcohol abuse
* Are taking medications or other substances contraindicated due to the nature of the study medication or the potential for drug interactions. This includes:

  * patients with allergies to prescription or OTC products containing NSAIDs
  * patients in whom aspirin or other NSAIDs or analgesic drugs induce the syndrome of asthma, rhinitis and nasal polyps
  * patients taking medications that may affect clotting, for example warfarin, parenteral heparin, ticlopidine (Ticlid®) or clopidogrel (Plavix®)
  * patients taking lithium
  * patients taking methotrexate
* Are renally or hepatically impaired in the judgment of the investigator based on the patient's medical history or other available clinical laboratory information
* Are taking sleep medications, muscle relaxants, anticonvulsants or antidepressants at a dose that has not been stable for at least 3 months
* Receiving physical therapy for the tendonitis/bursitis. Ongoing, stable physical therapy for conditions not related to tendonitis/bursitis is allowed.
* Have scheduled elective surgery or other invasive procedures during the period of study participation
* Have any illness or concurrent condition that would, in the opinion of the investigator or medical monitor, make study participation unsafe or would confound study results (e.g.,inflammatory arthritis, spondyloarthropathies, fibromyalgia, or are currently undergoing treatment for chronic pain)
* Have received an investigational drug or product or participated in an investigational drug study within a period of 30 days prior to receiving study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To measure the time to onset of action of the KTP in the treatment of pain associated with acute tendonitis or bursitis of the shoulder, elbow, or knee as measured by the time to meaningful pain relief. | 3 consecutive days

SECONDARY OUTCOMES:
Assess the safety and tolerability of the KTP as measured by adverse events cutaneous AEs, assessments of local tolerability and patch adherence, and vital signs | 3 consecutive days
Assess the time to first perceptible pain relief | 3 consecutive days
Assess the effect of KTP in the treatment of pain associated with acute tendonitis or bursitis of the shoulder, elbow or knee as measured by pain intensity during activity and pain relief. | 3 consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Endo Pharmaceuticals
Locations (2):
- United States (2):
  - HOPE Research Institute, LLC, Phoenix, Arizona
  - CPI, Clinical Research Atlanta, Stockbridge, Georgia